CLINICAL TRIAL: NCT04375995
Title: The Prevalence Of Small Airways Dysfunction In Asthma Patients And The Impact On The Asthma Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sibel Naycı (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Sibel Naycı, Prof. Dr., Mersin University
Organization: Mersin University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-2-TP3-3539-1
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Asthma; Small Airway Disease
Keywords: Asthma; Small Airway Dysfunction; Impulse oscillometry
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Fractional Exhaled Nitric Oxide Testing; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma group (Other): Impulse oscillometric pulmonary function tests and spirometric pulmonary function test will be performed to all asthmatic patients.To evaluate the degree of disease inflammation and phenotype, nitric oxide measurements will be made in the breath air with fractional exhaled nitric oxide (FENO) device. Blood eosinophil values will be examined. Thorax computed tomography will be performed to evaluate small airway dysfunction. Asthma control test (ACT) and asthma quality of life scale (AQLQ) will be applied. All patients will be followed for 1 year to record the number of exacerbations requiring emergency and hospital admissions for asthma.
  Interventions: Diagnostic Test: Impulse oscillometry; Diagnostic Test: Spirometric pulmonary function test; Diagnostic Test: Fractional exhaled nitric oxide (FENO) test; Diagnostic Test: Thorax Computed Tomography; Diagnostic Test: Blood eosinophil level; Other: Asthma control test; Other: Asthma quality of life scale
- Healthy control group (Other): Impulse oscillometric pulmonary function test, spirometric pulmonary function test and chest x ray will be performed.
  Interventions: Diagnostic Test: Impulse oscillometry; Diagnostic Test: Spirometric pulmonary function test; Diagnostic Test: Chest X Ray

INTERVENTIONS:
Diagnostic Test: Impulse oscillometry — Impulse oscillometry test will be applied to all groups.
Diagnostic Test: Spirometric pulmonary function test — Spirometric pulmonary function test will be applied to all groups.
Diagnostic Test: Fractional exhaled nitric oxide (FENO) test — FeNO test will be applied to asthma group.
  Arms: Asthma group
Diagnostic Test: Thorax Computed Tomography — Thorax Computed Tomography will be taken to the asthma group.
  Arms: Asthma group
Diagnostic Test: Blood eosinophil level — The blood eosinophil level will be evaluated to determine the phenotype in the asthma group.
  Arms: Asthma group
Other: Asthma control test — Asthma control test questions will be applied to the asthma group.
  Arms: Asthma group
Other: Asthma quality of life scale — Asthma quality of life scale (AQLQ) will be applied to the asthma group.
  Arms: Asthma group
Diagnostic Test: Chest X Ray — Chest X Ray will be applied to the healthy control group.
  Arms: Healthy control group

SUMMARY:
Asthma, which are one of the most important causes of morbidity and mortality both in the world and in our country, constitute a very serious social and economic burden. An estimated 300 million people suffer from asthma worldwide, which is a major public health problem. Asthma is complex and heterogeneous chronic airway diseases that require a multifaceted approach. In asthma, small airways represent key regions of airflow obstruction. Although small airway dysfunction is known in chronic airway diseases, the importance of small airway dysfunction on disease control, exacerbations and quality of life, and the importance of taking place among treatable targets is not clear. Thus, there is an unmet need to assess its role in the control of the disease. Therefore, our primary aim in the study is to determine the frequency of small airway dysfunction measured by impulse oscillometry in Asthma patients. Our secondary aim is to evaluate the role of small airway dysfunction in disease severity, disease phenotypes, disease control, quality of life and its effect on predicting the risk of exacerbation and its role among treatable targets in Asthma.

DETAILED DESCRIPTION:
This is a prospective cross-sectional interventional design. 73 asthmatic patients who applied to Mersin University Faculty of Medicine Hospital Chest Diseases Clinic between 01.10.2019-01.04.2020 will be taken. 35 healthy volunteers who were admitted to our clinic within the same date range will be taken as control group. Impulse oscillometric pulmonary function tests will be performed to all participants. Thorax computed tomography will be performed to evaluate small airway dysfunction. To evaluate the degree of disease inflammation and phenotype in asthma patients, nitric oxide measurements will be made in the breath air with fractional exhaled nitric oxide (FENO) device. The blood eosinophil level will be studied to determine the asthma phenotype.Asthma control test (ACT) will be applied to measure symptom control in patients with asthma. Asthma quality of life scale (AQLQ) will be applied to determine the quality of life in asthmatic patients. All patients will be followed for 1 year to record the number of exacerbations requiring emergency and hospital admissions for asthma. The effect of small airway dysfunction on asthma group, on the disease severity and control degree, disease phenotypes and quality of life, and the effect on the risk of exacerbation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Asthma group

* Participants who applied to the chest diseases clinic of Mersin University Hospital, between October 1, 2019 and April 1, 2020
* Participants who were diagnosed asthma with spirometry test
* Reading and signing Informed Consent Form
* Participants must be older than 18 years Healthy control group
* To apply to the chest diseases clinic of Mersin University Hospital between October 1, 2019 and April 1, 2020
* Reading and signing informed consent form
* Participants must be older than 18 years
* Must have no lung disease
* Must have no smoking history

Exclusion Criteria:

* Participants who do not sign the Informed Consent Form
* Under the age of 18 years
* Pregnant women
* Participants who with a history of cancer in the past 5 years
* Participants who previously had lung surgery
* Participants who with Interstitial Lung Disease
* Participants who with respiratory muscle disease
* Participants who with active pulmonary tuberculosis
* Participants who can not perform respiratory function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Small airway dysfunction will be evaluated by performing impulse oscillometry test. | through study completion, an average of 1 year
  We will used respiratory resistance at 5 and 20 Hz (R5 and R20, respectively) for the analyses. R5 and R20 are regarded as reflecting total and proximal airway resistance, respectively, and the fall in resistance from R5 to R20 (R5-R20) will used as a surrogate for the resistance of small airways.
Small airway dysfunction will be evaluated by thorax computed tomography. | through study completion, an average of 1 year
  Indirect changes caused by the small airways on the lung parenchyma will be detected by computed tomography (CT).
Small airway dysfunction will be evaluated by body plethysmography test. | through study completion, an average of 1 year
  Residual volume (RV) and total lung capacity (TLC) will be measured by body plethysmography test to determine small airway dysfunction.
Symptom control will be evaluated by asthma control test. | through study completion, an average of 1 year
  The asthma control test consists of 5 questions.
The number of moderate and severe exacerbations over a 1 year period will be recorded. | through study completion, an average of 1 year
  In the asthma group, each participant will be followed for 1 year in terms of recording exacerbations.
Forced expiratory volume in 1 second (fev1) change will be evaluated by spirometric pulmonary function test. | through study completion, an average of 1 year
  Forced expiratory volume in 1 second (fev1) change over one year period will be evaluated with spirometric pulmonary function test during recruitment and 1st year of follow-up.

SECONDARY OUTCOMES:
Quality of life will be evaluated by Asthma Quality of Life Questionnaire (AQLQ). | through study completion, an average of 1 year
  Asthma Quality of Life Questionnaire (AQLQ) contains 32 questions.
Fractional Exhaled Nitric Oxide (FENO) test will be used as an indicator of inflammation in determining the relationship between airway inflammation and small airway dysfunction. | through study completion, an average of 1 year
  FENO test is indirect measurements of inflammation, as used in clinical practice.
The relationship between blood inflammation cells and small airway dysfunction will be evaluated by complete blood count ( CBC). | through study completion, an average of 1 year
  Blood eosinophil and neutrophil levels will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Nayci, Prof.Dr., Study Chair — Mersin University, Department of Respiratory Diseases; Demet Polat Yulug, Dr., Principal Investigator — Mersin University, Department of Respiratory Diseases
Locations (1):
- Mersin University Faculty of Medicine, Department of Respiratory Diseases, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M; ATLANTIS study group. Exploring the relevance and extent of small airways dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med. 2019 May;7(5):402-416. doi: 10.1016/S2213-2600(19)30049-9. Epub 2019 Mar 12. PMID 30876830
- [Background] Usmani OS, Singh D, Spinola M, Bizzi A, Barnes PJ. The prevalence of small airways disease in adult asthma: A systematic literature review. Respir Med. 2016 Jul;116:19-27. doi: 10.1016/j.rmed.2016.05.006. Epub 2016 May 7. PMID 27296816